CLINICAL TRIAL: NCT00907088
Title: Nutritional Education and the Prevention of Iron Depletion in Children 9 Months to 2 Years: a Randomized Controlled Trial
Brief Title: Nutritional Education and the Prevention of Iron Depletion in Children 9 Months to 2 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Patricia Parkin, Staff Paediatrician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1000007781
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Iron Deficiency
Keywords: Iron depletion; Children; Educational intervention; Office-based
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Other: Standard nutrition counselling
- 2 (Experimental)
  Interventions: Other: Healthy milk intake

INTERVENTIONS:
Other: Healthy milk intake — In addition to the standard nutrition counselling, the intervention group will receive specific information regarding healthy milk intake (2 cups per day, maximum 16 ounces) and the potential negative health effects of prolonged bottle use and excessive milk intake including anemia, iron depletion, and dental carries.
  Arms: 2
Other: Standard nutrition counselling — Parents of children will receive nutrition counselling via trained study personnel, including recommendations for iron containing food choices and timing of cow's milk introduction. This group will also receive a colourful nutrition book.
  Arms: 1

SUMMARY:
Iron depletion in young children is common and may progress to iron deficiency anemia which is associated with irreversible neurodevelopmental effects. Efforts to prevent iron depletion are key to preventing these effects. In a recent study of 150 young children (12 to 38 months), we found that bottle fed children were almost three times as likely to be iron depleted compared with cup fed children (37% vs 18%). Thus, we hypothesize that an educational intervention designed to encourage timely bottle weaning will lead to a reduction in iron depletion.

DETAILED DESCRIPTION:
We plan to undertake a randomized controlled trial to evaluate the effectiveness of an office-based educational intervention for the prevention of iron depletion in young children. Healthy children will be recruited from a community pediatric office which serves a diverse, urban population. Children will be randomized to the intervention education group or the control education group at 9 months of age. Blood work (~4mL) for complete blood count and ferritin along with additional measures such as transferrin, iron, and reticulocyte count will be obtained at 24 months of age. Rates of iron depletion and anemia will be compared in the two groups. The two groups will also have 25-hydroxy vitamin D, calcium and alkaline phosphatase levels analyzed at the 24 month visit to ensure that the intervention for prevention of iron depletion does not adversely affect these measures.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9 months who are attending a routine primary care well-child visit.
* Children who are in good general health.
* Children whose parents provide informed consent to participate.

Exclusion Criteria:

* Children with chronic illness.
* Children with birth weight less than 2.5 kg.
* Children with previously diagnosed anemia (including known iron deficiency anemia). This includes children with marrow failure (aplastic anemia, Fanconi anemia), hemoglobinopathies (sickle cell disease, thalassemia), lead intoxication, sideroblastic anemia, megaloblastic anemia, enzymopathies (G6PD deficiency, pyruvate kinase deficiency), or membranopathies (hereditary spherocytosis).
* Children currently receiving medications associated with anemia. This includes children taking antimetabolites or phenytoin.
* Children currently receiving iron supplementation other than iron fortified formula.

Ages: 9 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Parkin, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Maguire JL, Birken CS, Jacobson S, Peer M, Taylor C, Khambalia A, Mekky M, Thorpe KE, Parkin P. Office-based intervention to reduce bottle use among toddlers: TARGet Kids! Pragmatic, randomized trial. Pediatrics. 2010 Aug;126(2):e343-50. doi: 10.1542/peds.2009-3583. Epub 2010 Jul 12. PMID 20624802

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Standard nutrition counselling: Parents of children will receive nutrition counselling via trained study personnel, including recommendations for iron containing food choices and timing of cow's milk introduction. This group will also receive a colourful nutrition book.
- Intervention Group: Healthy milk intake: In addition to the standard nutrition counselling, the intervention group will receive specific information regarding healthy milk intake (2 cups per day, maximum 16 ounces) and the potential negative health effects of prolonged bottle use and excessive milk intake including anemia, iron depletion, and dental carries.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 122 | 129
Completed | 102 | 99
Not Completed | 20 | 30

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Standard nutrition counselling: Parents of children will receive nutrition counselling via trained study personnel based on the Canadian Paediatric Society Guidelines. Nutrition counselling occurs at the 9-month visit and is repeated at the 15-month visit if the child has not transitioned into the use of a cup. Recommendations include iron containing food choices and timing of cow's milk introduction. This group will also receive a colourful nutrition book.
- Intervention Group: Healthy milk intake: In addition to the standard nutrition counselling provided in the control group, the intervention group will receive specific information regarding healthy milk intake (2 cups per day, maximum 16 ounces) and the potential negative health effects of prolonged bottle use and excessive milk intake including anemia, iron depletion, and dental carries.
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 122 | 129 | 251
Age, Categorical [Count of Participants; unit: Participants] — All participants were 9 months of age.
  Participants
    <=18 years | 122 | 129 | 251
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 66 | 119
  Male | 69 | 63 | 132
Race/Ethnicity, Customized [Number; unit: participants]
  White | 85 | 92 | 177
  Asian | 18 | 12 | 30
  Hispanic | 13 | 18 | 31
  Black | 6 | 7 | 13
Bottle use [Number; unit: participants]
  Breast Only | 46 | 38 | 84
  Bottle Only | 60 | 61 | 121
  Breast and Bottle | 15 | 26 | 41
  Information Not Available | 1 | 4 | 5
Plan to bottle-wean by 2 years old [Number; unit: participants]
  Plan to Bottle Wean By 2 Years Old | 67 | 63 | 130
  No Information Available | 55 | 66 | 121

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is Iron Depletion, and Will be Defined as Serum Ferritin <10 mcg/L.
Time Frame: Age 24 months
Measure: Number; unit: participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 99 | 102
participants
  No Iron Depletion | 64 | 71
  Yes Iron Depletion | 13 | 10
  Unknown | 22 | 21
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.42, Chi-squared

2. Secondary Outcome: Iron Deficiency (Defined as Serum Ferritin <10 mcg/L and MCV < 70 mcm3 Iron Deficiency.
Time Frame: Age 24 months
Reporting Status: Not Posted

3. Secondary Outcome: IDA (Hemoglobin < 110 g/L With Iron Deficiency)
Time Frame: Age 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/129
Other Adverse Events (participants affected / at risk) | 0/122 | 0/129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes